CLINICAL TRIAL: NCT00093041
Title: An Open, Single Dose Escalation Study Followed by a Multiple Dose Extension of Anti-EGF Receptor Human Monoclonal Antibody (Zalutumumab) in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Zalutumumab in Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hx-EGFr-001
Record Dates: First submitted 2004-09-30; First posted 2004-10-01 (Estimated); Results first posted 2011-12-22 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and neck cancer; squamous cell carcinoma of the head and neck
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — zalutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Zalutumumab 0.15 mg/kg (Experimental)
  Interventions: Drug: Zalutumumab
- Zalutumumab 0.5 mg/kg (Experimental)
  Interventions: Drug: Zalutumumab
- Zalutumumab 1 mg/kg (Experimental)
  Interventions: Drug: Zalutumumab
- Zalutumumab 2 mg/kg (Experimental)
  Interventions: Drug: Zalutumumab
- Zalutumumab 4 mg/kg (Experimental)
  Interventions: Drug: Zalutumumab
- Zalutumumab 8 mg/kg (Experimental)
  Interventions: Drug: Zalutumumab

INTERVENTIONS:
Drug: Zalutumumab — Weekly infusion
  Other Names: HuMax-EGFr

SUMMARY:
The purpose of this trial is to determine the safety of zalutumumab as a treatment for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of squamous cell carcinoma of the oral cavity, nasal cavity, paranasal sinuses, nasopharynx, oropharynx, hypopharynx or larynx.
* Primary or recurrent disease for which no curative or established palliative treatments are amenable
* WHO performance status of 1 or 2.

Exclusion Criteria:

* Received certain other treatments within 4 weeks prior to administration of study drug
* Previous severe allergic reactions (e.g. angio-edema, severe asthma, or anaphylaxis).
* Skin disease requiring systemic or local corticosteroid therapy.
* Known brain metastasis or leptomeningeal disease.
* Signs or symptoms of acute illness.
* Bacterial, fungal or viral infection.
* Certain serious medical conditions, including kidney or liver disease, some psychiatric illnesses, myocardial infarction within one year and stomach, lung, heart, hormonal, nerve or blood diseases.
* Pregnant or breast-feeding women.
* Women of childbearing age who are unable or unwilling to use an IUD or hormonal birth control during the whole trial.
* Simultaneous participation in any other trial involving investigational drugs or having participated in a trial within 4 weeks prior to start of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-12-01 (Actual); Primary Completion 2005-01-12 (Actual); Study Completion 2005-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (3):
  - Århus Kommunehospital, Århus C
  - Rigshospitalet, Copenhagen Ø
  - Odense Universitetshospital, Odense
- Sweden (2):
  - Universitets Sjukhuset i Lund, Lund
  - Uppsala Akademiska Sjukhus, Uppsala

REFERENCES:
- [Result] Bastholt L, Specht L, Jensen K, Brun E, Loft A, Petersen J, Kastberg H, Eriksen JG. Phase I/II clinical and pharmacokinetic study evaluating a fully human monoclonal antibody against EGFr (HuMax-EGFr) in patients with advanced squamous cell carcinoma of the head and neck. Radiother Oncol. 2007 Oct;85(1):24-8. doi: 10.1016/j.radonc.2007.06.007. Epub 2007 Jun 28. PMID 17602769

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zalutumumab 0.15 mg/kg | Zalutumumab 0.5 mg/kg | Zalutumumab 1 mg/kg | Zalutumumab 2 mg/kg | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Started | 4 | 4 | 5 | 4 | 4 | 7
Completed | 2 (One discontinued during single dose period and one during multiple dose period) | 1 (Three discontinued during single dose period) | 3 (Two discontinued during single dose period) | 3 (One discontinued during single dose period) | 3 (One discontinued during multiple dose period) | 4 (Three discontinued during multiple dose period)
Not Completed | 2 | 3 | 2 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zalutumumab 0.15 mg/kg | Zalutumumab 0.5 mg/kg | Zalutumumab 1 mg/kg | Zalutumumab 2 mg/kg | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg | Total
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 4 | 7 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 4 | 3 | 4 | 6 | 25
  >=65 years | 0 | 0 | 1 | 1 | 0 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] | 54 [49 to 62] | 59 [49 to 63] | 57 [56 to 68] | 55 [50 to 76] | 53 [47 to 61] | 58 [52 to 67] | 57 [47 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 0 | 1 | 6
  Male | 2 | 3 | 4 | 3 | 4 | 6 | 22
Region of Enrollment [Number; unit: participants]
  Denmark | 4 | 3 | 3 | 3 | 4 | 6 | 23
  Sweden | 0 | 1 | 2 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Number of participants reporting at least one adverse event.
Time Frame: From study start (Day 0) until follow-up period (up to Day 77)
Population: Number of participants reporting at least one adverse event
Measure: Number; unit: participants
Arm/Group | Zalatumumab 0.15 mg/kg | Zalutumumab 0.5 mg/kg | Zalutumumab 1 mg/kg | Zalutumumab 2 mg/kg | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 4 | 7
participants | 4 | 4 | 5 | 4 | 4 | 7

2. Secondary Outcome: Overall Response (OR), Classification
Description: Best Overall Response is defined as the best response from the start of treatment until disease progression (PD) /recurrence and was evaluated using Response Evaluation Criteria In Solid Tumors (RECIST). As per RECIST, PD is defined as at least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started, OR the appearance of one or more new lesions.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Zalatumumab 0.15 mg/kg | Zalutumumab 0.5 mg/kg | Zalutumumab 1 mg/kg | Zalutumumab 2 mg/kg | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 4 | 7
participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 1 | 0 | 1
  Stable Disease | 0 | 0 | 1 | 2 | 3 | 3
  Progression | 2 | 1 | 2 | 0 | 1 | 2
  Missing | 2 | 3 | 2 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: From study start (Day 0) until end of follow-up period (up to Day 77)
Arm/Group | Zalutumumab 0.15 mg/kg | Zalutumumab 0.5 mg/kg | Zalutumumab 1 mg/kg | Zalutumumab 2 mg/kg | Zalutumumab 4 mg/kg | Zalutumumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/4 | 3/4 | 5/5 | 1/4 | 0/4 | 6/7
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5 | 4/4 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 0.15 mg/kg (N=4) | Zalutumumab 0.5 mg/kg (N=4) | Zalutumumab 1 mg/kg (N=5) | Zalutumumab 2 mg/kg (N=4) | Zalutumumab 4 mg/kg (N=4) | Zalutumumab 8 mg/kg (N=7)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bleeding from tumour (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Administration site condition (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope vasovagal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zalutumumab 0.15 mg/kg (N=4) | Zalutumumab 0.5 mg/kg (N=4) | Zalutumumab 1 mg/kg (N=5) | Zalutumumab 2 mg/kg (N=4) | Zalutumumab 4 mg/kg (N=4) | Zalutumumab 8 mg/kg (N=7)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (5) | 5 (6)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 5 (6)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 4 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Headache (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Rigors (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 4 (5)
Sweating increased (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0)
Flushing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study comprised a single-dose escalation part for assessment of safety and a repeat dose extension including 4 weekly infusions. Please see the referred publication by Bastholt at al 2007 for detailed results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No